CLINICAL TRIAL: NCT05026684
Title: Achieving Greater Value for Veterans Through Full Cost Transparency
Brief Title: Value For Veterans (V4V)
Acronym: V4V
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: VA Ann Arbor Healthcare System (U.S. Federal Agency)
Collaborators: VA Center for Clinical Management Research (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: VAAnnArbor
Record Dates: First submitted 2021-08-09; First posted 2021-08-30 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Delivery of Health Care
Keywords: Cost; Value; Veterans; Behavioral Intervention; Personalized healthcare

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental): Personalized cost information group.
  Interventions: Other: Personalized cost handout

INTERVENTIONS:
Other: Personalized cost handout — Patients will be given a personalized cost handout to make transparent the full costs to Veterans of different types of ambulatory visits in order to optimize the value of their health care investments.

SUMMARY:
The COVID-19 pandemic has transformed the delivery of ambulatory care in the US. One of the most notable changes to ambulatory care practice has been the rapid expansion of telemedicine services. Such expansion sought to preserve access to necessary care for patients while protecting them and their clinicians from undue risk of exposure to COVID-19.

This multiphase, Veteran-centered approach to developing and evaluating a novel behavioral intervention to provide full cost transparency to Veterans will achieve the following aims:

Aim 1: Create an automated system to generate personalized estimates of Veterans' full costs (travel costs, time costs, and out-of-pocket costs) for different types of primary care visits.

Aim 2: Develop and refine a novel behavioral intervention that will help Veterans and their clinicians use personalized information about the full costs of different types of primary care visits in the VHA.

Aim 3: Evaluate the acceptability, feasibility, and preliminary effectiveness of the developed intervention to Veterans and their clinicians.

DETAILED DESCRIPTION:
Within VA Primary Care, the COVID-19 pandemic has resulted in an abrupt shift from mostly face-to-face visits to almost exclusively telephone and VA Video Connect (VVC) appointments. As the COVID-19 curve has flattened and personal protective equipment (PPE) supplies have stabilized, VA Medical Centers such as the VA Ann Arbor Healthcare System are now grappling with how to match these opportunities for different vehicles for delivering ambulatory care to patients' needs and preferences. One highly promising, Veteran-centered way to match opportunities for face-to-face, telephone, and VVC visits in the COVID-19 era is to consider the value each visit type yields for an individual Veteran. Value for a given health care service is broadly defined as its health outcomes (i.e., benefits) per dollars spent (i.e., costs). From the perspective of patients, costs entail not just out-of-pocket (OOP) expenses but also travel and time costs. These costs are even more salient for many Veterans in the current economic downturn which, unfortunately, is unlikely to abate until the US fully emerges from the COVID-19 pandemic. Careful consideration of these full costs -- which can vary widely across face-to-face, telephone, and VVC visits -- by both Veterans and their clinicians could result in higher-value ambulatory care visits. For example, when services could be provided by telephone rather than a face-to-face visit, the former would result in much higher value for Veterans because there are no copays or travel costs for telephone visits. Similarly, when a face-to-face visit is necessary, transparent cost information could encourage Veterans and their clinicians to maximize the necessary services delivered, amplifying the benefits realized for the relatively higher patient cost of that particular type of visit.

Despite the clear benefits of making patient costs more transparent, and of broader policy initiatives within VA to better inform Veterans' health care choices, Veterans and their clinicians currently lack the personalized cost information that they need to make high-value choices about ambulatory visit modalities. This project will make transparent the full costs to Veterans of different types of ambulatory visits in order to optimize the value of their health care investments in the COVID-19 era and beyond.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older with an upcoming face-to-face, telephone, or VVC appointment with a consenting Primary Care provider at the Ann Arbor VA.

Exclusion Criteria:

* Under the age of 18.
* Mild cognitive impairment, dementia, psychotic disorder, or unable to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-07-15 (Actual); Primary Completion 2022-05-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Level of confidence in understanding costs of different visit type options | Within one week of appointment
  Measured by telephone survey

SECONDARY OUTCOMES:
Conversations about different visit type options | Within one week of appointment
  Measured by telephone survey
Perceived helpfulness of intervention | Within one week of appointment
  Measured by telephone survey
Interest in receiving information in future | Within one week of appointment
  Measured by telephone survey

CONTACTS AND LOCATIONS:
Locations (1):
- VA Ann Arbor Healthcare System, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wosik J, Fudim M, Cameron B, Gellad ZF, Cho A, Phinney D, Curtis S, Roman M, Poon EG, Ferranti J, Katz JN, Tcheng J. Telehealth transformation: COVID-19 and the rise of virtual care. J Am Med Inform Assoc. 2020 Jun 1;27(6):957-962. doi: 10.1093/jamia/ocaa067. PMID 32311034
- [Background] Mann DM, Chen J, Chunara R, Testa PA, Nov O. COVID-19 transforms health care through telemedicine: Evidence from the field. J Am Med Inform Assoc. 2020 Jul 1;27(7):1132-1135. doi: 10.1093/jamia/ocaa072. PMID 32324855
- [Background] Porter ME. What is value in health care? N Engl J Med. 2010 Dec 23;363(26):2477-81. doi: 10.1056/NEJMp1011024. Epub 2010 Dec 8. No abstract available. PMID 21142528
- [Background] Farmer CM, Hosek SD, Adamson DM. Balancing Demand and Supply for Veterans' Health Care: A Summary of Three RAND Assessments Conducted Under the Veterans Choice Act. Rand Health Q. 2016 Jun 20;6(1):12. eCollection 2016 Jun 20. PMID 28083440
- [Background] Yabroff KR, Guy GP Jr, Ekwueme DU, McNeel T, Rozjabek HM, Dowling E, Li C, Virgo KS. Annual patient time costs associated with medical care among cancer survivors in the United States. Med Care. 2014 Jul;52(7):594-601. doi: 10.1097/MLR.0000000000000151. PMID 24926706
- [Background] Kullgren JT, Fagerlin A, Kerr EA. Completing the MISSION: a Blueprint for Helping Veterans Make the Most of New Choices. J Gen Intern Med. 2020 May;35(5):1567-1570. doi: 10.1007/s11606-019-05404-w. Epub 2019 Oct 24. PMID 31646457
- [Background] Department of Veterans Affairs FY 2018 - 2024 Strategic Plan. Published online February 12, 2018. Accessed April 10, 2018. https://www.va.gov/oei/docs/VA2018-2024strategicPlan.pdf
- [Background] Wait Times at Individual Facilities Search - VA Access to Care. Accessed May 2, 2018. https://www.accesstopwt.va.gov/
- [Background] How Does Your Medical Center Perform? Accessed May 2, 2018. https://www.va.gov/qualityofcare/apps/mcps-app.asp
- [Background] Final Report of the Commission on Care.; 2016. https://s3.amazonaws.com/sitesusa/wp-content/uploads/sites/912/2016/07/Commission-on-Care_Final-Report_063016_FOR-WEB.pdf
- [Background] John S. McCain III, Daniel K. Akaka, and Samuel R. Johnson VA Maintaining Internal Systems and Strengthening Integrated Outside Networks Act of 2018.; 2018. Accessed June 12, 2018. https://www.congress.gov/115/bills/s2372/BILLS-115s2372enr.xml
- [Background] Kullgren JT, Cliff EQ, Krenz C, West BT, Levy H, Fendrick AM, Fagerlin A. Consumer Behaviors Among Individuals Enrolled in High-Deductible Health Plans in the United States. JAMA Intern Med. 2018 Mar 1;178(3):424-426. doi: 10.1001/jamainternmed.2017.6622. PMID 29181512
- [Background] Kullgren JT, Cliff BQ, Krenz CD, Levy H, West B, Fendrick AM, So J, Fagerlin A. A Survey Of Americans With High-Deductible Health Plans Identifies Opportunities To Enhance Consumer Behaviors. Health Aff (Millwood). 2019 Mar;38(3):416-424. doi: 10.1377/hlthaff.2018.05018. PMID 30830816
- [Background] Kullgren JT. Helping Consumers Make High-Value Health Care Choices: The Devil Is in the Details. Health Serv Res. 2018 Aug;53 Suppl 1(Suppl Suppl 1):2655-2661. doi: 10.1111/1475-6773.12860. Epub 2018 Apr 16. No abstract available. PMID 29659010
- [Background] Thabane L, Ma J, Chu R, Cheng J, Ismaila A, Rios LP, Robson R, Thabane M, Giangregorio L, Goldsmith CH. A tutorial on pilot studies: the what, why and how. BMC Med Res Methodol. 2010 Jan 6;10:1. doi: 10.1186/1471-2288-10-1. PMID 20053272
- [Background] Kullgren JT, Krupka E, Schachter A, Linden A, Miller J, Acharya Y, Alford J, Duffy R, Adler-Milstein J. Precommitting to choose wisely about low-value services: a stepped wedge cluster randomised trial. BMJ Qual Saf. 2018 May;27(5):355-364. doi: 10.1136/bmjqs-2017-006699. Epub 2017 Oct 24. PMID 29066616
- [Background] Kullgren JT, Youles B, Shetty S, Richardson C, Fagerlin A, Heisler M. ForgIng New paths in DIabetes PrevenTion (FINDIT): Study Protocol for a Randomized Controlled Trial. Trials. 2017 Apr 8;18(1):167. doi: 10.1186/s13063-017-1887-6. PMID 28388933